CLINICAL TRIAL: NCT02783924
Title: The GLOBAL Vitamin D Study. A Genomic, Transcriptomic, Proteomic and Metabolomic Approach to the Effects of Vitamin D in Adipose Tissue and Peripheral Blood
Brief Title: The GLOBAL Vitamin D Study. A Genomic, Transcriptomic, Proteomic and Metabolomic Approach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: TromsøEndo-2012-2
Record Dates: First submitted 2016-04-22; First posted 2016-05-26 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2016-11

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; genomics; proteomics; metabolomics; adipose tissue
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecalciferol (Active Comparator): Vitamin d (as a 20.000 IU capsule) will be given i a dose of 40.000 IU per week for two months
  Interventions: Drug: Cholecalciferol
- Placebo (Placebo Comparator): two capsules (identical looking to the vitamin D capsules) will be given per week for two months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cholecalciferol — Vitamin D preparation
  Other Names: Dekristol
  Arms: Cholecalciferol
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
The effect of vitamin D supplementation on genetic, proteomic , and metabolomic profile in adipose tissue will be studied in 50 subjects.

DETAILED DESCRIPTION:
Vitamin D is a hormone with effects not only on the skeleton, but on most tissues in the body. Lack of vitamin D is associated with coronary heart disease, cancer and immunological diseases, and also with obesity, hypertension and glucose intolerance. However, to see the full effect of vitamin D, one should not only look at single diseases or risk factors, but have a global approach using a combined clinical index. A similar line of thinking can be applied to genetic, proteomic and metabolomic studies on vitamin D. Thus, in the present study 50 subjects will be included and randomized to vitamin D 40.000 IU per week versus placebo for 2 months. Blood and adipose tissue samples will be collected before and after the intervention and analyzed for gene expression. Based on these results the investigators will proceed with the relevant proteomic and metabolomic profile analyses. If successful, this may reveal new aspects of vitamin D's physiology and metabolic effects.

ELIGIBILITY:
Inclusion Criteria:

* serum 25OHD in the range 20 - 40 nmol/L
* no change in medication last 4 weeks

Exclusion Criteria:

* women < 60 yrs of age (to avoid influence of menstrual cycle)
* reduced kidney function
* serious diseases (cardio-vascular, diabetes, etc)
* taking vitamin d supplementation

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mRNA (messenger ribonucleic acid) profile in adipose tissue biopsies | 2 months

SECONDARY OUTCOMES:
Change from baseline in proteomic profile with relative quantification in adipose tissue biopsies with the use of Liquid chromatography mass spectrometry Technology (LC-MS/MS) | 2 months
Change from baseline in metabolomic profile with relative quantification in adipose tissue biopsies with the use of Liquid chromatography mass spectrometry Technology (LC-MS/MS) | 2 months
Effect of DBP (vitamin D binding protein) polymorphisms on the serum 25OHD response | 2 months
Effect of VDR (vitamin D receptor) polymorphisms on change from baseline in metabolomic profile with relative quantification in adipose tissue biopsies with the use of LC-MS/MS | 2 months
Effect of VDR (vitamin D receptor) polymorphisms on change from baseline in proteomic profile with relative quantification in adipose tissue biopsies with the use of LC-MS/MS | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: rolf Jorde, Professor, Principal Investigator — University of Tromso
Locations (1):
- university Hospital of North Norway, Tromsø, Norway

IPD SHARING:
Plan to Share IPD: No
not planned